CLINICAL TRIAL: NCT00131092
Title: Exercise Advice by Human or Computer: Testing 2 Theories
Brief Title: The CHAT (Community Health Advice by Telephone) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AG0033; R01AG016587 (NIH); Sponsored Proj. Office #20047
Record Dates: First submitted 2005-08-08; First posted 2005-08-17 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Health Behavior; Healthy
Keywords: exercise; aging; physical activity
MeSH Terms: conditions — Health Behavior; Motor Activity

INTERVENTIONS:
Behavioral: The Stanford Active Choices program
Behavioral: The TLC system

SUMMARY:
The purpose of the study is to compare a telephone-administered physical activity counseling program delivered by a person or by a telephone-linked computer system and test their relative benefits in improving regular physical activity among adults ages 55 and older.

DETAILED DESCRIPTION:
Two hundred and twenty five healthy, sedentary men and women ages 55 and older will be randomly assigned to one of three conditions: 12 months of physical activity counseling delivered by a human counselor, 12 months of physical activity counseling delivered by a telephone-linked computer system, or a 12-month attention-control condition (a health education class). Data on physical activity participation and related quality of life indicators (e.g., improved physical functioning, fitness, sleep) will be collected at baseline, 6 months, 12 month post-test and 18 month follow-up. The primary hypotheses are:

* participants in either physical activity counseling condition will show greater improvements in physical activity participation at 12 months compared to the attention-control condition;
* participants in the human counselor condition will show greater improvements in physical activity at 12 months relative to the computer condition; and
* participants in the computer condition will show better maintenance of physical activity between 12 and 18 months compared to participants in the human counselor condition.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 55 and older
* Free of any medical condition that would limit participation in independent exercise
* Not currently engaged in a regular pattern of physical conditioning
* Free of clinical psychopathology
* Stable on current medications
* Planning to remain in the geographic area through the duration of the trial
* Able to read and speak English sufficiently to understand protocol materials
* Can use the telephone unaided
* Willing to accept random assignment to any study condition

Exclusion Criteria:

* Under the age of 55
* Currently under treatment for an acute, serious medical condition (e.g., cancer, heart disease, stroke)
* Physically active on a regular basis (i.e. performing more than 60 minutes per week of aerobic physical activity of at least a moderate intensity)
* Unstable and/or uncontrolled on medications for high blood pressure or depression
* Unable or unwilling to use a telephone unaided
* Unwilling to accept random assignment to study condition

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225
Dates: Start 1999-06; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Increase in physical activity measured by the Stanford 7-Day Physical Activity Recall and the Community Healthy Activities Model Program for Seniors (CHAMPS) physical activity questionnaire for older adults

SECONDARY OUTCOMES:
Physical performance on a symptom-limited, graded exercise treadmill test
quality of life and psychological questionnaires measuring physical functioning, sleep, perceived stress, depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Abby C. King, PhD, Principal Investigator — Stanford Prevention Research Center
Locations (1):
- Stanford Prevention Research Center, Stanford, California, United States

REFERENCES:
- [Background] King AC, Friedman R, Marcus B, Castro C, Forsyth L, Napolitano M, Pinto B. Harnessing motivational forces in the promotion of physical activity: the Community Health Advice by Telephone (CHAT) project. Health Educ Res. 2002 Oct;17(5):627-36. doi: 10.1093/her/17.5.627. PMID 12408207
- [Background] Castro CM, King AC. Telephone-assisted counseling for physical activity. Exerc Sport Sci Rev. 2002 Apr;30(2):64-8. doi: 10.1097/00003677-200204000-00004. PMID 11991539
- [Background] Pinto BM, Friedman R, Marcus BH, Kelley H, Tennstedt S, Gillman MW. Effects of a computer-based, telephone-counseling system on physical activity. Am J Prev Med. 2002 Aug;23(2):113-20. doi: 10.1016/s0749-3797(02)00441-5. PMID 12121799
- [Background] Glanz K, Shigaki D, Farzanfar R, Pinto B, Kaplan B, Friedman RH. Participant reactions to a computerized telephone system for nutrition and exercise counseling. Patient Educ Couns. 2003 Feb;49(2):157-63. doi: 10.1016/s0738-3991(02)00076-9. PMID 12566210